CLINICAL TRIAL: NCT00552136
Title: Canadian Orthopaedic Foot and Ankle Society Surgical Treatment of Ankle Arthritis Outcome Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Orthopaedic Foot and Ankle Society (Other); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-MG-001
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Ankle Arthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Ankle; Replantation; Gene Fusion

ARMS (2):
- Ankle Arthroplasty (Active Comparator)
  Interventions: Procedure: Ankle Arthroplasty
- Ankle Artrodeses (Active Comparator)
  Interventions: Procedure: Ankle Arthrodesis

INTERVENTIONS:
Procedure: Ankle Arthroplasty
  Other Names: Replacement
  Arms: Ankle Arthroplasty
Procedure: Ankle Arthrodesis — Ankle fusion surgery
  Other Names: Fusion
  Arms: Ankle Artrodeses

SUMMARY:
The purpose of this study is to see if the clinical outcome success rate of Total Ankle Arthroplasty is similar to that of Ankle Arthrodesis over a period of 10 years. This will include looking at whether Total ankle arthroplasty results in a lower rate of hindfoot arthrosis and arthritis after surgery compared to ankle joint arthrodesis and if the rate of complications and revision surgery is acceptable when compared to Ankle Arthrodesis over a period of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) or older
* Known to have ankle arthritis for more than six (6) months
* Tried non operative treatment measures (eg. activity modification, physiotherapy, orthotics, bracing etc.) and have not improved
* Patient tests (questionnaires) show that ankle arthritis is severe
* Patient willing to take part in the study, including signing consent form after carefully reading it

Exclusion Criteria:

* Dead Bone in the Ankle
* Severe foot or Ankle Deformity
* Prior Ankle Fusion or Replacement
* Active or Prior Infection in the Ankle
* Obesity (greater than 250 lbs)
* Medical Conditions precluding safe surgery
* Nerve or Muscle disease
* Severe osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-05-30 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
AAOS Foot and Ankle Questionnaire - includes SF-36 | 10 years
AOFAS Ankle-Hindfoot Scale | 10 years
Ankle Osteoarthritis Scale | 10 years
Foot Function Index | 10 years
Radiographs | 10 years
Complications | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Glazebrook, MD, Principal Investigator — Capital District Health Authority, Halifax Canada; Tim Daniels, MD, Principal Investigator — St. Michael's Hospital (Toronto, Canada); Alistair Younger, MD, Principal Investigator — British Columbia Canada; Johnny Lau, MD, Principal Investigator — TorontoWestern Hospital, Toronto Canada; Peter Dryden, MD, Principal Investigator — Victoria, British Columbia Canada; Murry Penner, MD, Principal Investigator — British Columbia,Canada; Kevin Wing, MD, Principal Investigator — British Columbia, Canada; Craig Stone, MD, Principal Investigator — Newfoundland, Canada; Dave Stevens, MD, Principal Investigator — Waterloo, Ontario Canada
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada